CLINICAL TRIAL: NCT07390123
Title: A Randomized, Double-blind, and Placebo-controlled Parallel Phase Ⅲ Clinical Study to Evaluate the Efficacy and Safety of HSK39297 Tablets in Treatment of Patients With Primary IgAN
Brief Title: Phase Ⅲ Study of Efficacy and Safety of HSK39297 Tablet in Treatment of Patients With Primary IgAN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK39297-303
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: IgA Nephropathy (IgAN)
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- HSK39297 200mgQD (Experimental)
  Interventions: Drug: HSK39297

INTERVENTIONS:
Drug: HSK39297 — HSK39297 200mg, once a day; treatment period; 48-weeks fixed dose.
  Arms: HSK39297 200mgQD
Drug: Placebo — Placebo, once a day; treatment period; 48-weeks fixed dose.
  Arms: Placebo

SUMMARY:
Evaluate the efficacy and safety of HSK39297 tablets in patients with primary IgAN

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have signed and dated an IRB/IEC approved written informed consent form.Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, tumor biopsies, and other requirements of the study.
2. Female and male patients above 18 years of age.
3. Patients must weigh at least 35 kg to participate in the study, and must have a body mass index (BMI) below 35 kg/m2. BMI = Body weight (kg) / [Height (m)]2
4. Subjects with a biopsy-verified IgA nephropathy and where the biopsy was performed within the prior ten years.
5. 24h-UPCR ≥0.75g/g or 24h-UPE≥1.0g/24h at screening.
6. Measured Glomerular Filtration Rate (GFR) or estimated GFR (using the CKD-EPI formula 2021) ≥30 mL/min per 1.73 m2.For patients with eGFR* 20 to <30ml/min/1.73m2, a qualifying biopsy performed in two years.

Exclusion Criteria:

1. Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 90 days, whichever is longer.
2. All transplanted patients (any organ, including bone marrow).
3. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in-situ cervical cancer).
4. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study.
5. Pregnant or nursing (lactating) women.
6. Plasma donation (≥ 400mL) within 12 weeks prior to first dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Ratio to baseline in Urine Protein to Creatinine Ratio (sampled from 24h urine collection) at 36 weeks | From week 1 to week 36
Annualized total estimated Glomerular Filtration Rate slope over 48 weeks | From week 1 to week 48

SECONDARY OUTCOMES:
Annualized total estimated Glomerular Filtration Rate slope over 36 weeks | From week 1 to week 36
Annualized total estimated Glomerular Filtration Rate slope over 104 weeks | From week 1 to week 104
Incidence , severity and relationship of adverse events during the study period | From week 1 to week 108

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No